CLINICAL TRIAL: NCT04777773
Title: The Effect of Dual-task Training on Activity and Participation in Children With Cerebral Palsy
Brief Title: Dual-task Training in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sema BÜĞÜŞAN ORUÇ (Other)
Responsible Party: Sponsor-Investigator, Sema BÜĞÜŞAN ORUÇ, Research Assistant, Ordu University
Organization: Ordu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ordu347
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Palsy; Diplegia; Hemiplegic Cerebral Palsy; Physical Disability; Participation, Patient; Activity, Motor
Keywords: cerebral palsy; dual-task training; activity; participation
MeSH Terms: conditions — Cerebral Palsy; Patient Participation; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): classical physical therapy+ classical physical therapy
  Interventions: Other: dual-task training
- study group (Other): classical physical therapy+ dual-task training
  Interventions: Other: dual-task training

INTERVENTIONS:
Other: dual-task training — dual-task training

SUMMARY:
There are studies investigating the dual-task effect in sitting, standing up without sitting and walking in children with spastic CP. Some of these studies investigated motor-motor, some of them motor-cognitive dual-task states, and children with CP were compared to typically developing children. In all these studies, it is clearly seen that children with CP have more dual-task complexities than their typically developing peers. Some of these studies draw attention to dual-task education in children with CP. However, other than a randomized controlled study and a case report in the literature, we did not find any studies investigating the effectiveness of dual-task training in children with CP. When the literature is examined in detail, there is no study that examines the effect of dual-task exercise programs on walking activities and children's participation in daily life in children with CP.

This study has been planned based on this deficiency in the literature. Based on ICF, This study has been planned dual-task training for children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with cerebral palsy,
* Having spastic type unilateral and bilateral involvement,
* Being between the ages of 7-18,
* Being GMFCSS Level I and Level II,
* Continuing normal education (not being a mainstreaming student),
* Not having any surgical operation involving the musculoskeletal system in the last 6 months,
* Not having Botulinum Toxin application in the last 6 months.

Exclusion Criteria:

* Failing to accomplish the cognitive task (starting from a number between 0-100 and not counting back 1 each)
* Being a behavioral problem that makes it difficult to participate in the study,
* Inability to walk without support

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
10m walking test | 5 min
  10m walking test (the speed of gait is measured)
10m walking test with dual-task | 5 min
  10m walking test with dual-task (the speed of gait is measured) (dual- task is counting backwards)
10m backward walking test | 5 min
  10m backward walking test (the speed of gait is measured)
10m backward walking test with dual-task | 5 min
  10m backward walking test with dual-task (the speed of gait is measured) (dual- task is counting backwards)
balance | 15 min
  Balance skills of participators are assessed with 'Pediatric Berg Balance' .
participation of daily life | 15 min
  Participation of daily life of children are assessed with PODCI questionnaire.
Visual Gait Assessment | 10 min
  Participators' positions of joints are assessed with Edinburg Visual Score. Children walked 10m walking pathway. The camera records were frontside, backward, and laterals.

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu Uni, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No